CLINICAL TRIAL: NCT03126526
Title: Targeting Top-down and Bottom-up Processing in Eating Disorders Using Computerized Training Approaches: A Multimodal Outcome Study
Brief Title: A Multimodal Outcome Study of Eating Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Collaborators: University of Exeter (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRAS Project ID: 209609
Record Dates: First submitted 2017-04-03; First posted 2017-04-24 (Actual); Last update posted 2019-10-24 (Actual); Status verified 2019-10

CONDITIONS: Eating Disorder; Healthy
MeSH Terms: conditions — Feeding and Eating Disorders

STUDY DESIGN:
Intervention Model Description: The model includes two interventions (i.e. inhibitory control training and implementation intentions) that aim to target cognitive processes that have been reported to play a role in the onset and maintenance of eating disorders. Moreover, three arms exist, one for healthy controls including only one EEG assessment, and two interventional arms for participants with eating disorders. Participants in one interventional arm will receive food-specific inhibitory control training, while participants in the other interventional arm will receive general inhibitory control training. These are delivered through a website task (go/no-go training),
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Food specific inhibitory control training (Experimental): The stimuli in this task will involve pictures of food.
  Interventions: Behavioral: Food specific Inhibitory control training; Behavioral: Implementation intentions
- General inhibitory control training (Active Comparator): The stimuli in this task will not involve pictures of food, but pictures of stationary and household items.
  Interventions: Behavioral: Implementation intentions; Behavioral: General inhibitory control training
- Baseline brain activation assessment (healthy controls) (No Intervention): This arm is included to assess brain activation using EEG among healthy controls at baseline in order to compare responses to participants with eating disorders.

INTERVENTIONS:
Behavioral: Food specific Inhibitory control training — It involves a go/no-go task in which participants are requested to respond by clicking a particular button when a specific stimulus appears and requested to withhold their response when another particular stimulus appears. Stimuli in this intervention include photos of food and non-food.
  Arms: Food specific inhibitory control training
Behavioral: Implementation intentions — It involves designing "if-then" strategies of behaviour. Participants will be asked to describe situations in which they feel they are more prone to behave in a way that is not congruent to their long term goals, and then to plan strategies to behave differently when faced with this situation in the future.
  Arms: Food specific inhibitory control training; General inhibitory control training
Behavioral: General inhibitory control training — It involves a go/no-go task in which participants are requested to respond by clicking a particular button when a specific stimulus appears and requested to withhold their response when another particular stimulus appears. Stimuli in this intervention include only non-food pictures.
  Arms: General inhibitory control training

SUMMARY:
This research project aims to explore the effectiveness of combined go/no-go training and implementation intentions in targeting binge eating frequency among people with binge eating disorder and bulimia nervosa.

The full intervention is 4 weeks long and consists of completing the training and food diaries every day and meeting with the researcher twice for EEG recording. Moreover, it involves completing questionnaires at baseline, at intervention completion, and one month after the intervention.

Moreover, healthy control participants will be recruitment to complete baseline questionnaires and take part in one EEG recording session in order to assess baseline differences in brain activation in response to computer tasks.

DETAILED DESCRIPTION:
Participants will learn about the study through flyers, e-mail, and social media (i.e. twitter and Facebook) which will describe the interventional nature of the study, the main eligibility criteria, and the researcher's contact information. Interested individuals will be asked to contact the researchers, who will then send an information sheet detailing the study procedure and what participation would involve. After reading the information sheet, interested individuals will be contacted by the researchers in order to confirm all eligibility criteria including diagnostic assessment. If these are met a PDF of the consent form will be sent to the participants, including information about their rights as participants and their ability to withdraw at any time without having to give a reason. Participants who sign the consent form will respond to the email with the attached document. Next, researchers will contact the participant to set an appointment to enter the lab for the first EEG recording. Before entering the lab, participants will be asked to complete a food diary and complete the complete a battery of questionnaires. The questionnaires include: 1) a demographic questionnaire, 2) eating disorders examination questionnaire, 3) food ratings test, 4) self-regulation of eating behaviour questionnaire for adults, 5) The negative urgency scale, 6) the adults eating behaviour questionnaire, 7) GAD-7, and 8) PHQ-9.

Upon participants' arrival to the lab, participants will be asked to complete the food rating task. Next, they will learn to complete the training tasks (i.e. food specific go/no-go and general go/no-go) and perform them during EEG recording. They will be offered the opportunity to ask questions relating to the task or the EEG at any time. Their weight will also be measured.

Participants will be asked to complete the training and complete food diaries every day for four weeks. The successful/ unsuccessful attempts at implementation intentions will be assessed weekly by a mentor. A researcher/clinician will discuss setting the implementation intention goals with the participant over email. At the end of the training, participants will enter the lab to re-complete the four tasks while researchers record brain activation using the EEG. They will also be asked to complete the food rating task again and their weight will be re-assessed. Before leaving, they will be asked to complete a feedback sheet in which they can express their experience with the training, in terms of facilitators and barriers and visual analogue scales that will ask participants to rate the acceptability, usefulness and level of burden experienced with training.

Participants will then be followed up at 1 month post-intervention; they will be asked to complete the battery of questionnaires used at baseline and post-intervention.

ELIGIBILITY:
Inclusion Criteria:

1) Diagnosis of an Eating Disorder (Bulimia Nervosa or Binge Eating Disorder); 2) No severe psychiatric comorbidity (e.g. psychosis); 3) Fluency in English; 4) No visual impairment; 5) No cognitive/neurological impairment; 6) No drugs or alcohol abuse; 7) No use of weight-loss medication; 8 No metabolic disorder; 9) Above 18 years old and below 60 years old.

Exclusion Criteria:

1) No diagnosis of an eating disorder; 2) Severe psychiatric comorbidity; 3) No English language fluency; 4) Visual impairment (not correctable with eye-wear); 5) Cognitive/neurological impairment; 6) Drug or alcohol abuse; 7) Use of weight-loss medication; 8) A metabolic disorder; 9) Below 18 years old and above 60 years old.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2017-11-26 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-06-01 (Actual)

PRIMARY OUTCOMES:
Change in eating disorder symptomatology | This will be assessed at baseline, intervention completion, and follow-up (1 month later)
  Decrease in binge eating frequency and decrease in compensatory behaviours.

SECONDARY OUTCOMES:
Change in weight/BMI | This will be assessed at baseline (Time 0), intervention completion (4 weeks), and follow-up (8 weeks)
  Weight will be measured by the researcher and BMI will be calculated.
Change in inhibitory control | This will be assessed at baseline (Time 0) and intervention completion (4 weeks).
  This will be assessed using the self-report measure of disinhibition and using the go/no-go computerized task.
Change in anxiety and depression symptoms | This will be assessed at baseline (Time 0), intervention completion (4 weeks), and follow-up (8 weeks)
  This will be assessed using the GAD and PHQ measures.
Changes in High Calorie Food Valuation | This will be assessed at baseline (Time 0) and post-intervention (4 weeks).
  This will be assessed using the food rating task.
Changes in Low Calorie Food Valuation | This will be assessed at baseline (Time 0) and post-intervention (4 weeks).
  This will be assessed using the food rating task.

CONTACTS AND LOCATIONS:
Overall Officials: Rayane Chami, MSc/ PhD Student, Principal Investigator — King's College London; Dr Valentina Cardi, PhD, Study Director — King's College London; Professor Janet Treasure, Study Director — King's College London; Dr Grainne McLoughlin, Study Director — King's College London
Locations (1):
- Eating Disorders Unit, Institute of Psychiatry, Psychology, and Neuroscience, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lowe MR, Friedman MI, Mattes R, Kopyt D, Gayda C. Comparison of verbal and pictorial measures of hunger during fasting in normal weight and obese subjects. Obes Res. 2000 Nov;8(8):566-74. doi: 10.1038/oby.2000.73. PMID 11156432
- [Background] Hunot C, Fildes A, Croker H, Llewellyn CH, Wardle J, Beeken RJ. Appetitive traits and relationships with BMI in adults: Development of the Adult Eating Behaviour Questionnaire. Appetite. 2016 Oct 1;105:356-63. doi: 10.1016/j.appet.2016.05.024. Epub 2016 May 20. PMID 27215837
- [Background] Whiteside, S. P., & Lynam, D. R. (2001). The Five Factor Model and impulsivity: Using a structural model of personality to understand impulsivity. Personality and Individual Differences, 30(4), 669-689. http://dx.doi.org/10.1016/S0191-8869(00)00064-7.
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Fairburn, C. G. (2008). Cognitive behavior therapy and eating disorders. Guilford Press
- [Background] Kliemann N, Beeken RJ, Wardle J, Johnson F. Development and validation of the Self-Regulation of Eating Behaviour Questionnaire for adults. Int J Behav Nutr Phys Act. 2016 Aug 2;13:87. doi: 10.1186/s12966-016-0414-6. PMID 27484457